CLINICAL TRIAL: NCT01589276
Title: Risk Factors and Results of Emergency Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: FH08
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emergency hernia repairs
- Elective hernia repairs

SUMMARY:
The aim of present study was to evaluate the clinical course after emergency ventral hernia repair in terms of 30-day-readmission, -reoperation and -mortality and to identify risk factors for emergency repair.

DETAILED DESCRIPTION:
All incisional, umbilical and epigastric hernias registered in the Danish Ventral Hernia Database

ELIGIBILITY:
Inclusion Criteria:

* All incisional, umblilical and epigastric hernia repiars

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hernia repairs registered in the Danish Ventral Hernia Database during the study period
Sampling Method: Non-Probability Sample
Enrollment: 10976 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
risk factors for emergency ventral hernia repair | 4 years
  evaluation of risk factors (hernia size, hernia type, type of surgery, age and gender) for poor outcome after emergency ventral hernia repair.

SECONDARY OUTCOMES:
30-day readmission | 30 days
  evaluation of risk factors (hernia size, hernia type, type of surgery, age and gender) for 30-day readmission after emergency ventral hernia repair
30-day reoperation | 30 day
  evaluation of risk factors (hernia size, hernia type, type of surgery, age and gender) for 30-day reaoperation after emergency ventral hernia repair
30-day mortality | 30 day
  evaluation of risk factors (hernia size, hernia type, type of surgery, age and gender) for 30-day mortality after emergency ventral hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — dept. surgery, Køge sygehus, Denmark
Locations (1):
- Dept. of Surgery, Køge Hospital, Køge, Denmark

REFERENCES:
- [Derived] Helgstrand F, Rosenberg J, Kehlet H, Bisgaard T. Outcomes after emergency versus elective ventral hernia repair: a prospective nationwide study. World J Surg. 2013 Oct;37(10):2273-9. doi: 10.1007/s00268-013-2123-5. PMID 23756775